CLINICAL TRIAL: NCT02906969
Title: Educational Colonoscopy Video Enhances Bowel Preparation Quality and Comprehension in an Inner City Population
Brief Title: Colonoscopy Educational Video Upon Inner City Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 1203000992
Record Dates: First submitted 2016-06-13; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Other Surgical Procedures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colonoscopy educational Video (Experimental): Brief educational video of colonoscopy to determine comprehension and quality of bowel preparation.
  Interventions: Other: Colonoscopy Educational Video
- Control (Placebo Comparator): Non-colonoscopy video as a control.
  Interventions: Other: Placebo Educational Video

INTERVENTIONS:
Other: Colonoscopy Educational Video — Brief Video utilization to assess comprehension and evaluation bowel preparation quality
  Arms: Colonoscopy educational Video
Other: Placebo Educational Video — Brief Video utilization to provide placebo information and evaluation bowel preparation quality
  Arms: Control

SUMMARY:
Background:

The investigators assessed the use of a colonoscopy instructional video to improve both bowel preparation and education prior to procedure. Preceding studies have been vague, pinning patient education via diagrams and text as both pivotal and useless for compliance in bowel preparations. These studies however lacked assessment of comprehension prior to procedure.

Methodology:

This is a prospective study of diverse, inner city outpatient university center, first time colonoscopy patients given 1 of 2 on-site videos and written/verbal instruction. Experimentals saw a 5 min video on the purpose of colonoscopy, bowel preparation, pre-colonoscopy diet, and proper laxative use. Controls saw a 5 min video from the same spokesperson on upper endoscopy; which was trivial. Both groups were given a quiz within 30 days of the colonoscopy on demographics, and 14 test questions about colonoscopy and preparation. Subsequently, endoscopists used the additive Ottawa scale to rate quality of preparation (range 0-14) via: fluid (0=sm,1=mod, 2=lg) and cleanliness in each the right, mid and rectosigmoid colon, (0=excellent, 1=good, 2=fair, 3=poor, 4=inadequate).

ELIGIBILITY:
Exclusion Criteria:

* Patients were excluded if they had dementia or
* cognitive impairment or
* if they did not have a pre-procedural office visit.

Inclusion Criteria:

* age 18-85
* undergoing initial outpatient colonoscopy
* willing to participate in and sign consent for this study
* Morning session of colonoscopy procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Primary outcome improvement in adequate bowel preparations | in 30 days retention from the video
  Bowel preparation quality indicator using Ottawa bowel prep scale.
Comprehension of colonoscopy/colorectal cancer screening | in 30 days retention from the video
  Questionnaire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rex DK, Imperiale TF, Latinovich DR, Bratcher LL. Impact of bowel preparation on efficiency and cost of colonoscopy. Am J Gastroenterol. 2002 Jul;97(7):1696-700. doi: 10.1111/j.1572-0241.2002.05827.x. PMID 12135020
- [Background] Spiegel BM, Talley J, Shekelle P, Agarwal N, Snyder B, Bolus R, Kurzbard N, Chan M, Ho A, Kaneshiro M, Cordasco K, Cohen H. Development and validation of a novel patient educational booklet to enhance colonoscopy preparation. Am J Gastroenterol. 2011 May;106(5):875-83. doi: 10.1038/ajg.2011.75. Epub 2011 Apr 12. PMID 21483463
- [Derived] Pillai A, Menon R, Oustecky D, Ahmad A. Educational Colonoscopy Video Enhances Bowel Preparation Quality and Comprehension in an Inner City Population. J Clin Gastroenterol. 2018 Jul;52(6):515-518. doi: 10.1097/MCG.0000000000000893. PMID 28742732